CLINICAL TRIAL: NCT01951807
Title: Psychological Interventions for Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 130909; R01CA085566-06A1 (NIH); NCI-2012-00551 (Other: CTRP (Clinical Trails Reporting Program))
Record Dates: First submitted 2013-05-07; First posted 2013-09-27 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Gynecologic Cancer
Keywords: Psychosocial Effects of Cancer and Treatment; Coping
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coping & Communication Skills (Experimental): The CCI intervention focuses on bolstering stress management and problem solving abilities, identifying and expressing support needs constructively, facilitating the ability to cope with unchangeable issues, cognitive restructuring, and dealing effectively with body image and sexuality issues over seven weekly 60 minute sessions.
  Interventions: Behavioral: Psychotherapy
- Supportive Counseling (SC) (Experimental): The SC intervention incorporates a supportive, non-directive counseling approach in seven weekly 60 minute sessions
  Interventions: Behavioral: Psychotherapy
- Usual Care (UC) (No Intervention): Patients receive standard psychological and emotional care (usual care [UC]) (i.e., social work consultations and referral to a psychiatrist or psychologist, if requested or deemed necessary by the attending physician).

INTERVENTIONS:
Behavioral: Psychotherapy
  Arms: Coping & Communication Skills; Supportive Counseling (SC)

SUMMARY:
Subjects that have received medical treatment for ovarian cancer can be both physically and emotionally demanding for patients. The purpose of this study is to determine whether two common pyschological interventions (Communication Skills Intervention and Supportive Counseling) may improve the well-being of ovarian cancer patients compared to usual care.

DETAILED DESCRIPTION:
Very little is known in the psycho-oncology literature about why psychological interventions are effective or for how long these interventions exert an impact. Given many cancer patients experience recurrence and/or progression, it is important to know whether our relatively brief interventions facilitate how patients cope with this most-feared medical event. From a theoretical perspective, the study will advance our understanding of the mechanisms for change for two common treatment approaches, supportive and cognitive behavioral therapies.

Subjects will be enrolled and upon completion of a baseline survey, randomized to into one of three arms - Communication Skills Intervention, Supportive Counseling, and Usual Care. Subjects will complete surveys during the course of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with any stage of primary ovarian cancer, primary peritoneal cancer, or primary fallopian tube cancer in the past 6 months
* Newly diagnosed with High Grade Stage 2, any grade Stage 3 or higher endometrial cancer in the past 6 months
* Newly diagnosed with Stage 2 or higher cervical cancer withing the past 6 months
* Newly diagnosed with any stage of Uterine cancer (both sarcoma and carcinosarcoma) in the past 6 months
* At the time of recruitment, the patient is on active treatment defined as either currently receiving chemotherapy or radiation or less than 6 months post-cancer surgery
* At the time of recruitment, a Karnofsky Performance Status of 80 or above or an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* English speaking
* Lives within a two-hour commuting distance from the recruitment site
* No hearing impairment
* Has signed consent within 6 months of diagnosis date

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2010-06; Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Do the two psychological interventions, CCI and SC, result in greater improvements in global psychological adaptation | 7 years
  Global Psychological distress:
  Depressive symptoms - The BDI is a 21-item scale which has been widely used in studies incorporating cognitive-behavioral interventions.The MHI-18 has subscales for Psychological Distress and Well-being.
Do the two psychological interventions, CCI and SC, result in greater improvements in cancer-specific psychological adaptation | 7 years
  Cancer-Specific Distress:
  Traumatic Stress. The Impact of Events Scale (IES) is a 15-item self-report measure focusing on intrusive and avoidant ideation related to gynecologic cancer and its treatment. Using a 4-point Likert scale, participants rated how true each statement has been for them during the past week (scale range = 0-75).
  Fear of Recurrence/Progression. The Concerns about Recurrence Scale (CARS) is a 26 item assessment of the nature of women's fears about cancer recurrence.
Do the two psychological interventions, CCI and SC, result in greater improvements in quality of life | 7 years
  Quality of Life-General. The Functional Assessment of Cancer Therapy - General (FACT-G) is a widely used measure of QOL. The FACT-G is comprised of 27 questions that assess well-being in four domains: physical, functional, social/family, and emotional.
  Spiritual well-being. The FACIT Spiritual well-being scale assesses a sense of meaning in life, harmony, peacefulness, sense of strength, and comfort from one's faith. The 12 item scale has two factors: Meaning/Peace and Faith.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Cooper Health System, Camden, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Jefferson University School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania